CLINICAL TRIAL: NCT05965180
Title: Interstitial Assessment of Architectural Heterogeneity in Prostate Cancer Using a Fine Needle Photoacoustic Probe
Status: Recruiting | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: UMCC 2022.015; HUM00217834 (Other: University of Michigan); R37CA222829 (NIH)
Record Dates: First submitted 2023-04-27; First posted 2023-07-28 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: Biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Biopsy: Patients will be identified once prostate biopsies have been scheduled. Once enrolled on trial, patients will undergo standard biopsy procedure as per clinical care. During this biopsy, research measurements will be completed using the fine needle photoacoustic probe.
  Interventions: Device: Fine Needle Photoacoustic Probe

INTERVENTIONS:
Device: Fine Needle Photoacoustic Probe — Fine Needle Photoacoustic Probe guided by the standard biopsy system without tissue core extraction

SUMMARY:
In this project, we will integrate the Photoacoustic (PA) technology into a prostate biopsy procedure through a fine needle probe. The needle probe will be in the shape of a biopsy needle and compatible with the needle insertion mechanism in the transrectal ultrasound (TRUS) probe. When inserted into the prostate, the fine needle PA probe will assess the histological information in its surrounding tissue without any tissue extraction. The needle probe has been tested in prostate tissue samples and whole human prostates ex vivo.

DETAILED DESCRIPTION:
14AUG2024- enrollment was increased to 50 subjects

ELIGIBILITY:
Inclusion Criteria:

* 1) Planned prostate biopsy as part of routine clinical care
* 2) > 40 and <80 years old

Exclusion Criteria:

* 1) Known history of bleeding disorders or
* 2) Patients taking anticoagulants, no matter doses or washout time
* 3) Known allergy to silicone material
* 4) Unable to provide informed consent
* 5) Either the surgeon or the patient do not think the patient will not be able to complete all parts of the study, the patient will be excluded
* 6) Involved in other investigational studies.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with planned prostate biopsy procedures will be recruited through U-M Urology Clinics
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Demonstration of reliable measurements | day 1
  The primary aim of this study is to demonstrate that our fine needle PA probe can acquire reliable measurements of prostate glands. This will be indicated by a signal-to-noise ratio of the measurements that is larger than one.
  We will calculate the signal to noise ratio of the signals as the peak-to-peak signal magnitude over the amplitude of the system background signal. The technical failure is that we will not be able to achieve measurements with signal-to-noise ratios larger than 1 in 10% of the measurements. We will have a futility analysis after first 5 patients are completed (thus 10 measurements). If of those 10 measurements, 2 have a SNR less 1, then the study will be stopped as it is unlikely to meet its 90% target.

SECONDARY OUTCOMES:
Determining the ability to observe differences between benign and cancerous regions | day 1
  The secondary aim of this study is documenting our ability to observe differences between the PASA linear slope values derived from benign and cancerous regions, i.e., to detect the difference of 0.05 of 0.19, 0.17, 0.14, 0.20 dB/MHz between the means of the linear slopes in benign and cancerous regions at the wavelengths of 1220 nm, 1370 nm, 800 nm and 266 nm, respectively.
  We will aim at differentiating the measurements in benign and cancerous regions at specific wavelengths. We have a null hypothesis for each wavelength that at this specific wavelength, our measurement cannot differentiate the benign and cancerous regions. We will test the hypothesis with paired t-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Guan Xu, Phd, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No